CLINICAL TRIAL: NCT06712732
Title: Valutazione Ultrasonografica Del Corretto Posizionamento Della Maschera Laringea Nel Paziente Pediatrico
Brief Title: Ultrasound Evaluation of Laryngeal Mask Airway (LMA) Placement in Pediatric Patients and Its Relationship to Postoperative Complications
Acronym: LMAUSPED
Status: Not yet recruiting | Type: Observational
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Rachele Simonte, Medical Doctor, Researcher, University Of Perugia
Other Study IDs: LMAUSPED
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Paediatric Airway

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was designed to improve understanding of some respiratory reactions that can occur after surgery, such as difficulty breathing or persistent cough. These events, technically called PRAE (postoperative respiratory complications), are common reactions in children who have undergone surgery, and our aim is to find out if there are signs that can help us predict them, reducing their incidence in the future.

During surgery, the child will receive general anesthesia, which will put him or her to sleep and not feel pain. In this context, a laryngeal mask airway (LMA) will be used to help the child breathe. The laryngeal mask airway is a soft device that is placed in the throat and allows the airway to be kept open, making breathing possible. This is a standard tool that will be used during surgery regardless of participation in the study.

The aim of this study is to better understand the relationship between the correct positioning of the laryngeal mask airway, measured by a specific ultrasound score, and the frequency of postoperative respiratory events in pediatric patients. As previously stated, these complications are common and well known in pediatric anesthesia practice, and the study aims to explore whether adequate ultrasound assessment can help predict and prevent them in the future. The study aims to observe the position of the laryngeal mask airway through a simple ultrasound and verify whether there is a relationship between the way the mask is positioned and the possibility of postoperative respiratory events. This type of ultrasound is non-invasive and does not add risk to the child.

This ultrasound check will take place without affecting the normal treatment of the patient and does not involve any additional risk or discomfort.

The study is purely observational: this means that we will collect information without modifying in any way the care already foreseen for the child.

The laryngeal mask airway and neck ultrasound are already part of standard medical practice, and the study does not present any additional risks. In this case, it is only a matter of reporting in all children who will participate in the study the "results" of ecological story of the neck (which we will process according to a score) and to evaluate whether there is a relationship between this score and the occurrence of respiratory adverse events upon awakening.

The overall duration of the study is 24 months. In total, we expect to include about 340 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery under general anesthesia with laryngeal mask airway placement.

Exclusion Criteria:

* Patients without the need for invasive airway management or undergoing surgery requiring orotracheal intubation.
* Patients with known craniofacial malformations.
* Patients undergoing neck surgery.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients undergoing surgery under general anesthesia with laryngeal mask airway placement.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation between PRAE incidence and correlation with ultrasound score | From enrollment to the discharge from the recovery room
  The aim of this observational study is to evaluate whether there is a correlation between ultrasonographic data and the incidence of postoperative complications in pediatric patients undergoing general anesthesia for surgery, in order to evaluate the possible predictive power on complications of this diagnostic technique. Postoperative complications or PRAE (Perioperative Respiratory Adverse Events) are: major complications (bronchospasm and laryngospasm) and minor complications (desaturation <95%, signs of airway obstruction with increased effort of accessory respiratory muscles and/or snoring, severe cough for more than 10s continuously, postoperative stridor, presence of blood traces at removal of the LMA)